CLINICAL TRIAL: NCT06555289
Title: Visual and Refractive Outcomes of the Clareon PanOptix Pro IOL in Patients With Prior Myopic Refractive Surgery
Brief Title: Outcomes of Clareon PanOptix Pro in Patients With Prior Myopic Refractive Surgery
Status: Recruiting | Type: Observational
Sponsor: Juliette Eye Institute Research Center (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Other Study IDs: RM-24-01
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Clareon PanOptix Pro IOL — Spherical and toric T3

SUMMARY:
This study is a Single center, single arm, prospective, observational study of clinical outcomes following bilateral cataract surgery and Clareon PanOptix Pro implantation. Subjects will be assessed preoperatively, and at 1 and 3 months postoperatively. Clinical evaluations will include administration of the QUVID and IOLSAT questionnaires, manifest refraction, topography, as well as measurement of visual acuities at distance, intermediate, and near.

ELIGIBILITY:
Inclusion Criteria:

* Adults (45 years or older) who have confirmed age-related cataracts and are eligible for bilateral cataract surgery.
* Prior binocular myopic photorefractive keratectomy (PRK) or myopic LASIK.
* Patients who have regular corneal astigmatism less than or equal to 0.6 D and are candidates for the PanOptix Pro spherical IOL.
* Patients who have regular corneal astigmatism and are candidates for PanOptix Pro toric IOL T3
* Postoperative visual potential of monocular 20/25 or better, in the surgeon's judgement.

Exclusion Criteria:

* Any ocular comorbidity that might hamper postoperative visual acuity:

  * Corneal abnormality including corneal dystrophy, irregularity, and degeneration.
  * Moderate or severe dry eyes that can't be relieved after treatment.
  * History of or current anterior and posterior inflammation of any etiology.
  * Retinal pathology such as AMD, diabetic retinopathy, vein occlusion, etc.
  * Glaucoma of any kind.
  * Pregnancy or lactation.
* Any ocular surgery other than corneal myopic refractive surgery (LASIK and PRK).
* Patients with physical or intellectual disability (e.g. Down's Syndrome, Parkinson's Disease, unable to fixate)
* Apple Kappa/chord mu ≥ 0.6.
* Higher order corneal aberrations at pupil diameter of 4mm: > 0.6 total RMS, > 0.3 coma, > 0.3 trefoil (to exclude irregular corneas)
* Any patient requiring a limbal relaxing incision.

The principal investigator reserves the right to declare a patient ineligible or non-evaluable based on medical evidence that indicates they are unsuitable for the trial.

Min Age: 45 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Eligible test subjects will be those with age-related cataracts and prior myopic refractive surgery.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Binocular corrected distance visual acuity (logMAR) | 3 months postoperative

SECONDARY OUTCOMES:
Binocular distance corrected visual acuity at intermediate (logMAR) | 3 months postoperative
Binocular distance corrected visual acuity at near (logMAR) | 3 months postoperative
Binocular unccorrected visual acuity at distance (logMAR) | 3 months postoperative
Binocular unccorrected visual acuity at intermediate (logMAR) | 3 months postoperative
Binocular unccorrected visual acuity at near (logMAR) | 3 months postoperative

OTHER OUTCOMES:
Visual Disturbance Questionnaire | 3 months postoperative
  Questionnaire for Visual Disturbances (QUVID). Lower scores indicate less frequent, severe, or bothersome visual disturbances.
Satisfaction Questionnaire | 3 months postoperative
  The Intraocular Lens Satisfaction questionnaire (IOLSAT). Lower scores indicate higher spectacle independence and satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Melendez, MD, MBA, Principal Investigator — Juliette Eye Institute Research Center
Locations (1):
- Juliette Eye Institute Research Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No